CLINICAL TRIAL: NCT02130453
Title: Use of Regadenoson for a Stress Echocardiogram Protocol Using Speckle Tracking Imaging
Brief Title: Accuracy of an Echo-Stress Protocol Using Regadenoson With Speckle Tracking
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Astellas Scientific & Medical Affairs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2013-0881; NCI-2014-01162 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Results first posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-07

CONDITIONS: Ischemia
Keywords: Ischemia; Coronary artery disease; Nuclear stress test; Stress Echocardiogram; Echocardiography strain measurement; Ultrasound cardiac imaging; ReSTE; SPECT; Regadenoson
MeSH Terms: conditions — Ischemia; Coronary Artery Disease | interventions — regadenoson

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ReSTE Cardiac Imaging (Experimental): Echocardiography strain measurement performed taking about 10 minutes. After resting strain measurement done, first set of nuclear images performed. Once these images are completed, participant given Regadenoson 0.4 mg by vein over about 10 seconds. Within 2 to 4 minutes of receiving the Regadenoson, measurements repeated. These measurements will take about 2 minutes to complete.
  Interventions: Drug: Regadenoson
- SPECT Cardiac Imaging (Other): After resting strain measurement done, first set of nuclear images taken. Once these images are completed, participant given Regadenoson 0.4 mg by vein over about 10 seconds. Within 2 to 4 minutes of receiving Regadenoson, measurements repeated. These measurements take about 2 minutes to complete. At about 30 minutes after Regadenoson given, participant will have final images for the nuclear portion of the testing.
  Interventions: Drug: Regadenoson

INTERVENTIONS:
Drug: Regadenoson — 0.4 mg by vein given during nuclear stress testing with echocardiography strain measurements.

SUMMARY:
The goal of this clinical research study is to compare regadenoson nuclear stress testing with echocardiography strain measurements (an ultrasound imaging method that measures hearts function) in detecting coronary artery disease.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will have the echocardiography strain measurement performed. This will be done while you lie on an exam table. An ultrasound technician will apply a vaseline-like gel to your chest and will take the measurements by holding a transducer (a device that resembles a microphone) against your chest, sliding it back and forth. This will take about 10 minutes.

After the resting strain measurement is done, you will have the first set of nuclear images. This will be done just like the echocardiography strain measurement. Once these images are completed, you will be given regadenoson by vein over about 10 seconds. Within 2 to 4 minutes of receiving the regadenoson, measurements will be repeated. These measurements will take about 2 minutes to complete. At about 30 minutes after regadenoson was given, you will have the final images for the nuclear portion of the testing (this is the usual timing for nuclear images after regadenoson).

You will receive the same treatment during your stress test, including the same amount of regadenoson, as you would if you did not take part in this study. Some participants may be asked to allow a repeat of the strain measurements that will include an additional dose of regadenoson if the first set of images are not good enough and additional images may be taken.

Length of Study:

Your participation on this study will be over 30 days after the tests OR after surgery, whichever occurs later. Researchers will collect information from your medical record for up to 30 days after your tests.

If you have surgery or are hospitalized in the 30 days after the tests, you will be called and asked about any problems you have been having. This call should take about 10 minutes.

This is an investigational study. Regadenoson is FDA approved and is routinely used for nuclear perfusion stress testing. The use of strain measurement during an echocardiogram to detect coronary disease is investigational.

Up to 300 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients who are scheduled for (perfusion) nuclear stress testing using regadenoson as stress agent.
2. Indications for stress testing is either: -as part of a pre-operative evaluation prior to a planned cancer related surgery that is considered to be at least of intermediate risk (Intra-peritoneal, intra-thoracic, head and neck surgery, orthopedic or prostate surgery) OR -as an evaluation in the cardiology clinic for symptoms described in a cardiology consult as typical angina, or of significant suspicion for coronary disease or symptoms described as likely of a cardiac/coronary etiology.
3. Patients with a history of LV dysfunction will be still candidates for enrollment in the study if they have documented LVEF recovery (most recent documented LVEF of 50% or higher) for at least 6 months prior to SPECT regardless of current cardiac medication regimen.
4. Age 18 - 80 years.

Exclusion Criteria:

1. Patients consented for the trial that on the baseline 2D study have poor acoustic echo windows (i.e. a reader is unable to see in definition 2 or more segments from the apical views) will not be eligible to continue in the trial and peak hyperemia images will not be obtained.
2. Any patient with tachycardia defined as HR of 100 or higher at the day of SPECT will not be eligible for this study.
3. Second- or third- degree AV block.
4. Sinus node dysfunction.
5. Patients with allergy to regadenoson.
6. Patients with LBBB and/or artificial pacemaker.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas L Palaskas, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the cardiac stress laboratory at MD Anderson's main building between 9-30-2014 and 9-7-2018. Patients who were scheduled for a nuclear stress test using regadenoson were evaluated for eligibility and approached for participation in the study.
Pre-assignment Details: 161 participants were approached for the study but 27 participants were excluded. The reasons for exclusion prior to inclusion in the study were as follows: poor quality echocardiographic images (24 patients), patient withdrew consent (2 patients), surgery canceled (1 patient)
Groups:
- Experimental: ReSTE Cardiac Imaging: Echocardiography strain measurement performed taking about 10 minutes. After resting strain measurement done, first set of nuclear images performed. Once these images are completed, participant given Regadenoson 0.4 mg by vein over about 10 seconds. Within 2 to 4 minutes of receiving the Regadenoson, measurements repeated. These measurements will take about 2 minutes to complete.
Period: Overall Study
Arm/Group | Experimental: ReSTE Cardiac Imaging
Started | 134
Completed | 134
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: ReSTE Cardiac Imaging
Number analyzed (Participants) | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.99 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 117
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 111
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 134

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Accuracy of ReSTE Imaging to SPECT Imaging in Diagnosis of Ischemia
Description: As primary analysis, paired test of equivalence used for proportions proposed by Tango to test equivalence of the two ischemia tests among tSPECT positive patients.
Time Frame: 1 day
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Experimental: ReSTE Cardiac Imaging
Number analyzed (Participants) | 134
proportion of participants
  Positive RESTE proportion with positive angiogram | 0.1538 [0.0151 to 0.2925]
  Positive nuclear stress test proportion with positive angiogram | 0.2308 [0.0688 to 0.3928]

2. Secondary Outcome: Cardiac Event Rates After ReSTE and SPECT Imaging
Description: Cardiac events after ReSTE and SPECT imaging included myocardial infarction,heart failure, sudden cardiac death, cerebrovascular accident
Time Frame: 30 days
Population: Evaluation of cardiac events within 30 days of surgery for those patients who had SPECT for preoperative evaluation.
Measure: Number; unit: events
Arm/Group | Experimental: ReSTE Cardiac Imaging
Number analyzed (Participants) | 68
events | 0

ADVERSE EVENTS:
Time Frame: 30 days after surgery
Arm/Group | Experimental: ReSTE Cardiac Imaging
All-Cause Mortality (participants affected / at risk) | 0/134
Serious Adverse Events (participants affected / at risk) | 0/134
Other Adverse Events (participants affected / at risk) | 0/134

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT02130453/Prot_SAP_000.pdf